CLINICAL TRIAL: NCT06682273
Title: The Combination of Thread-embedding and Auricular Acupuncture in the Treatment of Non-specific Chronic Low Back Pain
Brief Title: Thread-embedding Combined With Auricular Acupuncture for Non-specific Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Tin Trong Nguyen, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 273HDDD-GD
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Chronic Non-Specific Low Back Pain
Keywords: acupuncture; thread embedding acupuncture; auricular acupuncture; low back pain; traditional medicine
MeSH Terms: conditions — Low Back Pain | interventions — Acupuncture, Ear

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TEA + AA (Experimental): Thread-embedding acupuncture (TEA) every week in 4 weeks (4 sessions). Combined with auricular acupuncture (AA) every week in 4 weeks (4 sessions).
  Interventions: Other: Thread-embedding acupuncture; Other: Auricular acupuncture
- TEA + sham AA (Active Comparator): Thread-embedding acupuncture (TEA) every week in 4 weeks (4 sessions). Combined with sham auricular acupuncture (sham AA) every week in 4 weeks (4 sessions).
  Interventions: Other: Thread-embedding acupuncture; Other: Sham auricular acupuncture
- AA + sham TEA (Active Comparator): Auricular acupuncture (AA) every week in 4 weeks (4 sessions). Combined with sham thread-embedding acupuncture (sham TEA) every week in 4 weeks (4 sessions).
  Interventions: Other: Auricular acupuncture; Other: Sham thread-embedding acupuncture
- Sham both (Sham Comparator): Sham thread-embedding acupuncture (sham TEA) every week in 4 weeks (4 sessions). Combined with sham auricular acupuncture (sham AA) every week in 4 weeks (4 sessions).
  Interventions: Other: Sham thread-embedding acupuncture; Other: Sham auricular acupuncture

INTERVENTIONS:
Other: Thread-embedding acupuncture — Thread-embedding acupuncture is performed every week for 4 weeks, using a single Polydioxaone thread inserted into acupoints on the body through the needle. After the thread is inserted, the needle will be immediately withdrawn.
  Arms: TEA + AA; TEA + sham AA
Other: Auricular acupuncture — Auricular acupuncture is conducted weekly for 4 weeks using patches, each with a square shape and a side length of 10 mm, along with a sterilized needle measuring 0.25 x 1.3 mm inserted into therapeutic points on the ear. The patches with the needle will remain in place for one week.
  Arms: AA + sham TEA; TEA + AA
Other: Sham thread-embedding acupuncture — Sham thread-embedding acupuncture is performed every week for 4 weeks, using the needle without thread inserted into acupoints on the body. After insertion, the needle will be immediately withdrawn, and no thread will be left in the body.
  Arms: AA + sham TEA; Sham both
Other: Sham auricular acupuncture — Sham auricular acupuncture is conducted weekly for 4 weeks using patches, each with a square shape and a side length of 10 mm, along with a sterilized needle measuring 0.25 x 1.3 mm inserted into non-therapeutic points on the ear. The patches with the needle will remain in place for one week.
  Arms: Sham both; TEA + sham AA

SUMMARY:
Low back pain (LBP) is a significant global health issue, with cases expected to rise by 36.4% by 2050. Chronic LBP (cLBP), lasting over three months, is mostly non-specific cLBP (cNLBP), posing a challenge for effective management. Common treatments include medication, exercise, and acupuncture.

This study explores the combined use of thread-embedding and auricular acupuncture for treating cNLBP, as combining these methods is thought to enhance effectiveness. Participants with cNLBP will be randomized into four groups to receive either the combination of both treatments, each treatment individually with a sham, or both shams. The study will last eight weeks, with four weeks of intervention and four weeks of follow-up. Treatment outcomes, including pain, disability, medication use, and quality of life, will be evaluated, along with monitoring for adverse effects.

DETAILED DESCRIPTION:
Low back pain (LBP) is a major public health issue worldwide. In 2020, there were over half a billion cases of LBP globally, and by 2050, the total number of LBP cases is expected to increase by 36.4% worldwide. LBP accounts for 7.7% of total Years Lived with Disability, making it the largest contributor to the global disability burden.

When lasting three months or more, LBP is classified as chronic (cLBP). Most cLBP is non-specific cLBP (cNLBP). Managing cNLBP remains challenging. Recommended therapies include short-term medication, manipulation, supervised exercise, cognitive behavioral therapy, and multidisciplinary treatment. According to the Clinical Practice Guideline from the American College of Physicians, clinicians and patients should initially consider non-pharmacologic treatments, including acupuncture as one of the options.

There is evidence regarding the effectiveness of thread-embedding acupuncture (TEA) and auricular acupuncture (AA) in the treatment of cNLBP. TEA uses the principle of selecting points on the body, while AA involves selecting points on the ear. The difference in the point selection principles of these two methods has led clinicians to often combine them in hopes of enhancing treatment efficacy. However, evidence on the effectiveness of combining these two methods in treating cNLBP remains lacking. This study aims to clarify whether the combination of these methods is more effective than using them individually.

Eligible participants with cNLBP, defined as LBP lasting more than three months without any reasonable explanation and determined by a physician to be nonspecific, will be enrolled and subsequently randomized into four groups: receiving the combination of TEA and AA (TEA + AA group), receiving TEA and sham AA (TEA + sham AA group), receiving AA and sham TEA (AA + sham TEA group), and receiving sham TEA and sham AA (Sham both group), with a 1:1:1:1 allocation ratio.

The study will last for eight weeks, with four weeks of intervention and four weeks of follow-up. AA and sham AA will be administered weekly during the four-week intervention (four sessions). TEA and sham TEA will be administered every two weeks during the four-week intervention (two sessions). Data on treatment efficacy will include disability index, pain score, amount of analgesic medication needed, quality of life score, and global improvement. Additionally, adverse effects will be monitored and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with low back pain at the outpatient clinic.
* Diagnosed with non-specific low back pain persisting for more than 3 months, without radiation to the legs.
* Pain-NRS score ≥ 4 on a 10-point scale.
* Independent ambulation capability (with or without walking aids).
* Consent to participate in the study.

Exclusion Criteria:

* History of prior lumbar spine surgery.
* Known or suspected severe spinal conditions (e.g., cancer, vertebral fracture, spinal infection, or cauda equina syndrome).
* Signs of concurrent involvement of lumbar nerve roots, plexus, sciatic nerve, other leg nerves, or diagnosed polyneuropathy confirmed by electrodiagnosis.
* Presence of systemic inflammatory diseases, including rheumatoid arthritis, gout, ankylosing spondylitis, or psoriatic arthritis.
* Unstable or untreated severe health conditions (such as end-stage renal disease, advanced liver failure, NYHA class IV heart failure).
* Alcohol abuse or substance dependence.
* Use of anti-inflammatory medication within 2 weeks prior to enrollment.
* Acupuncture treatment within the past 4 weeks.
* Previous treatment with thread-embedding or auricular acupuncture for any condition.
* Damaged skin in the acupuncture area or history of hypersensitivity reactions to acupuncture.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index (ODI) percentage score | Week 0, Week 2, Week 4, Week 6, and Week 8
  The Oswestry Disability Index (ODI) percentage score evaluates the impact of low back pain on various activities (sleeping, self-care, sex life, social life, and traveling) using six rating options (0 to 5). Participants select the most appropriate response, and the total score is calculated as a percentage of the maximum possible score (50 if all sections are completed). A score of zero indicates no disability, while a score of 100% implies significant disability.

SECONDARY OUTCOMES:
Change in pain score on the Numeric Rating Scale (NRS) | Week 0, Week 2, Week 4, Week 6, and Week 8
  The pain score on the Numeric Rating Scale (NRS) is a subjective measure used to assess the intensity of pain experienced by an individual. Participants are asked to rate their pain on a scale from 0 to 10, where 0 represents no pain and 10 indicates the worst possible pain.
Change in the number of paracetamol tablets used | Week 2, Week 4, Week 6, and Week 8
  The number of paracetamol 500mg tablets used per week will be recorded.
Change in the Patient-Reported Outcomes Measurement Information System Global Health 10 (PROMIS-GH-10) score | Week 0, Week 2, Week 4, Week 6, and Week 8
  The Patient-Reported Outcomes Measurement Information System Global Health 10 (PROMIS-GH-10) is a 10-item assessment tool that includes ratings for four general items (health, quality of life, physical health, and mental health) and six additional items covering five health domains: physical function (1 item), fatigue (1 item), pain (1 item), emotional distress (1 item), and social health (2 items). Each question has five response options ranging from 1 to 5, except for the pain scale, which ranges from 0 to 10. The total score ranges from 9 to 55, with higher scores indicating better quality of life.
Global improvement rate | Week 2, Week 4, Week 6, and Week 8
  Global improvement is assessed through the patients global impression of change, using a 7-point scale: 1 = completely recovered, 2 = greatly improved, 3 = somewhat improved, 4 = no change, 5 = somewhat worse, 6 = significantly worse, and 7 = extremely worsened. Participants who score 1 or 2 are considered improved, those with scores of 3 to 5 are classified as unchanged, and scores of 6 or 7 indicate deterioration.
Proportion of intervention-related adverse events | Up to eight weeks
  For thread-embedding acupuncture and sham thread-embedding acupuncture, anticipated adverse events include local discomfort, an increase in body temperature following treatment, local hematoma or subcutaneous bleeding, local swelling, induration, pain, redness, infection, abscess, itching, and anaphylaxis. Anticipated adverse events for auricular acupuncture and sham auricular acupuncture include pain at the insertion site, local discomfort, skin irritation (itching and redness), local inflammation and bleeding, chondritis, dizziness, nausea, and hypersensitivity reactions. Additionally, any unforeseen adverse events related to these procedures are documented and monitored.

CONTACTS AND LOCATIONS:
Locations (1):
- Nhan Dan Gia Dinh Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hunter RF, McDonough SM, Bradbury I, Liddle SD, Walsh DM, Dhamija S, Glasgow P, Gormley G, McCann SM, Park J, Hurley DA, Delitto A, Baxter GD. Exercise and Auricular Acupuncture for Chronic Low-back Pain: A Feasibility Randomized-controlled Trial. Clin J Pain. 2012 Mar-Apr;28(3):259-67. doi: 10.1097/AJP.0b013e3182274018. PMID 21753728
- [Background] Lee HJ, Choi BI, Jun S, Park MS, Oh SJ, Lee JH, Gong HM, Kim JS, Lee YJ, Jung SY, Han CH. Efficacy and safety of thread embedding acupuncture for chronic low back pain: a randomized controlled pilot trial. Trials. 2018 Dec 12;19(1):680. doi: 10.1186/s13063-018-3049-x. PMID 30541604
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Maughan EF, Lewis JS. Outcome measures in chronic low back pain. Eur Spine J. 2010 Sep;19(9):1484-94. doi: 10.1007/s00586-010-1353-6. Epub 2010 Apr 17. PMID 20397032
- [Background] Haefeli M, Elfering A. Pain assessment. Eur Spine J. 2006 Jan;15 Suppl 1(Suppl 1):S17-24. doi: 10.1007/s00586-005-1044-x. Epub 2005 Dec 1. PMID 16320034
- [Derived] Pham TL, Le NT, Nguyen TT, Chu H. Should thread-embedding and auricular acupuncture be combined rather than used individually for non-specific chronic low back pain?: A double-blinded, randomized, sham-controlled trial. Integr Med Res. 2025 Sep;14(3):101180. doi: 10.1016/j.imr.2025.101180. Epub 2025 Jun 13. PMID 40689022